CLINICAL TRIAL: NCT01063491
Title: Cardiac CAtheterization for Bypass Graft Patency Rate Optimization: the CABG-PRO Randomized-controlled Pilot Study
Acronym: CABG-PRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Director, Cardiac Catheterization Laboratories, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-001
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Bypass Graft Surgery
Keywords: coronary artery bypass graft surgery; bypass grafts; angiography; percutaneous coronary intervention; coronary imaging; coronary artery bypass graft surgery, bypass graft patency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early graft angiography after coronary artery bypass surgery (Experimental): Treatment of any bypass graft abnormalities that are discovered will be performed if needed
  Interventions: Procedure: bypass graft angiography
- No early angiography after coronary artery bypass surgery (No Intervention)

INTERVENTIONS:
Procedure: bypass graft angiography
  Arms: Early graft angiography after coronary artery bypass surgery

SUMMARY:
Aortocoronary bypass graft failure is common and is associated with high morbidity and mortality. Failure of saphenous vein grafts is more common than failure of internal mammary artery grafts. Whether early graft angiography can reduce bypass graft failure remains unknown. The Cardiac CAtheterization for Bypass Graft Patency Rate Optimization (CABG-PRO) randomized-controlled pilot study is a phase III, double-blind, randomized-controlled pilot trial that will randomize 170 patients undergoing coronary artery bypass graft surgery to early (before dismissal) graft angiography vs. no early graft angiography. Coronary angiography will be performed at 12 months, to determine whether compared to no early graft angiography, early graft angiography will result in:

1. lower per patient angiographic bypass graft failure (in at least one graft) rates (defined as ≥75% diameter stenosis in at least one bypass graft) (primary efficacy endpoint)
2. lower per graft failure rates, per graft occlusion rates, and per patient bypass graft occlusion rates (in at least one bypass graft) (secondary endpoints)
3. lower incidence major adverse cardiac events (death, nonfatal myocardial infarction, nonfatal stroke, coronary revascularization, and composite of death/myocardial infarction) (secondary endpoint)

Intravascular ultrasonography and near-infrared spectroscopy will also be performed in at least one bypass graft at baseline (in the early graft angiography group only) and at 12-month angiographic follow-up to evaluate the structural bypass graft changes occurring after coronary artery bypass graft surgery (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Willing and able to give informed consent. The patients must be able to comply with study procedures and follow-up.
3. Undergoing clinically-indicated coronary artery bypass graft surgery

Exclusion Criteria:

1. Positive pregnancy test or breast-feeding
2. Coexisting conditions that limit life expectancy to less than 12 months or that could affect a patient's compliance with the protocol
3. Serum creatinine > 2.5 mg/dL or acute renal failure
4. Severe peripheral arterial disease limiting vascular access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Per patient bypass graft failure (defined as ≥75% graft diameter stenosis) in at least one bypass graft, as assessed by quantitative coronary angiography performed at 12 months. | 12 months

SECONDARY OUTCOMES:
Per graft incidence of bypass graft failure; per graft incidence of bypass graft occlusion; and per patient incidence of at least one bypass graft occlusion | 12 months
Major adverse cardiac events (death, nonfatal myocardial infarction, nonfatal stroke, coronary revascularization, and composite of death/myocardial infarction) | 12 months
Mean SVG lumen diameter and wall thickness, as assessed by intravascular ultrasonography and mean lipid core burden index, as assessed by near-infrared intracoronary spectroscopy | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- VA North Texas Healthcare System, Dallas, Texas, United States